CLINICAL TRIAL: NCT00384813
Title: Project ASPIRE: Improving Pediatric Asthma Management for Urban Families
Brief Title: Family-Focused, Stress-Reduction Program to Improve the Health Care of Urban Children With Asthma
Acronym: ASPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marianne Celano, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 014-2006; R21HL083877 (NIH); 014-2006 (Other: Emory IRB)
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Home-based family intervention (Experimental): Home-based family intervention
  Interventions: Behavioral: Project ASPIRE Home-Based Family Intervention
- 2: ETAU (Active Comparator): Enhanced Treatment As Usual (1 home visit)
  Interventions: Behavioral: Project ASPIRE Enhanced Treatment As Usual

INTERVENTIONS:
Behavioral: Project ASPIRE Home-Based Family Intervention — Home-based psychoeducational family intervention jointly conducted by psychology postdoctoral fellow and respiratory therapist over 4 months
  Arms: 1: Home-based family intervention
Behavioral: Project ASPIRE Enhanced Treatment As Usual — Psychoeducational family intervention addressing the written asthma action plan during a single home visit, conducted by a respiratory therapist
  Arms: 2: ETAU

SUMMARY:
Stress and anxiety can negatively affect children with asthma. Reducing the stress of asthmatic children and their families may lead to improved asthma care and fewer asthma symptoms in the children. The purpose of this study is to develop and evaluate a family-focused asthma education program aimed at reducing stress levels and improving asthma care for urban children with asthma.

DETAILED DESCRIPTION:
Asthma is a serious, chronic illness that affects 9 million children in the United States. Common asthma symptoms include wheezing, shortness of breath, chest tightness, and coughing. Asthma attacks can be triggered by a variety of irritants, including mold, pollen, tobacco smoke, or allergies. Stress can also cause asthma attacks, and children who experience high levels of stress and anxiety tend to have poor asthma management skills and health outcomes. Additionally, family stress can affect the ability of families and caregivers to provide adequate care to children with asthma. Currently, few asthma education programs are aimed at helping both children and parents manage stress. The purpose of this study is to evaluate the effectiveness of a stress-reduction family intervention on improving health outcomes in asthmatic children.

Study researchers will first conduct focus groups with children who have asthma, their parents, and community health organizations to identify barriers to effective asthma management and sources of stress for caregivers; a family-focused intervention will then be developed. Fifty families with an asthmatic child will be enrolled and randomly assigned to one of two groups. Group 1 participants will partake in four to six home-based, family educational sessions over a 4-month period. Sessions will focus on asthma education and stress management techniques for the entire family. One of these sessions may take place at the child's doctor's office as a way to focus on improving parent-doctor communication. Group 2 participants will partake in a single home-based asthma education session. Study visits for all participants will occur at baseline, Month 4, and 6 months post-intervention. At these timepoints, asthma self-management will be assessed through family interviews and observation of the child's inhaler use; tobacco exposure levels will be measured with a urine test; and family functioning and stress levels will be assessed with questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of persistent asthma
* Poorly controlled asthma, as determined by emergency department visit, hospitalization, or steroid burst in the year prior to study entry
* Primary caregiver is under stress, as determined by a significantly elevated score on measures of stress
* Receives Medicaid or participates in Medicaid HMO
* Resides in the Atlanta metropolitan area

Exclusion Criteria:

* Nonatopic, nonpsychiatric illness that requires daily medication
* Diagnosis of asthma in the year prior to study entry
* Homeless
* Caregiver is unable to complete study screening process
* Caregiver does not speak English

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2007-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marianne P. Celano, PhD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University School of Medicine, Atlanta, Georgia
  - American Lung Association - Southeast Division, Smyrna, Georgia

REFERENCES:
- [Result] Celano MP, Holsey CN, Kobrynski LJ. Home-based family intervention for low-income children with asthma: a randomized controlled pilot study. J Fam Psychol. 2012 Apr;26(2):171-8. doi: 10.1037/a0027218. Epub 2012 Feb 20. PMID 22353006

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Families were recruited from an urban hospital and a residential camp for children with asthma. Initial eligibility criteria : (a) residence in one of two urban counties, (b) child age 8 to 13, (c) Medicaid or State Children's Health Insurance Program, (d) current prescription of a daily controller agent, and (e) poorly controlled asthma.
Pre-assignment Details: Caregivers of children meeting initial eligibility criteria were interviewed briefly by phone; those answering affirmatively to either of two stress questions were invited to participate in a Screening Assessment. Caregivers with an elevated score on a stress measure were invited to participate in the trial.
Groups:
- 1: Home-based Family Intervention: Home-based family intervention
  Project ASPIRE Home-Based Family Intervention : Home-based psychoeducational family intervention jointly conducted by psychology postdoctoral fellow and respiratory therapist over 4 months
- 2: Enhanced Treatment As Usual: Enhanced Treatment As Usual (1 home visit)
  Project ASPIRE Enhanced Treatment As Usual : Psychoeducational family intervention addressing the written asthma action plan during a single home visit, conducted by a respiratory therapist
Period: Overall Study
Arm/Group | 1: Home-based Family Intervention | 2: Enhanced Treatment As Usual
Started | 23 | 20
Completed | 21 | 20
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1: Home-based Family Intervention | 2: Enhanced Treatment As Usual | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (1.4) | 10.6 (1.9) | 10.5 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15
  Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 19 | 40
  White | 0 | 0 | 0
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Score on the Family Asthma Management System Scale (FAMSS)
Description: Family Asthma Management System Scale is semi-structured clinical interview that includes open-ended questions assessing family management of pediatric asthma. The interview is recorded and rated using a standard manual on seven core subscales and two optional subscales.The interview is recorded and rated on seven to nine 9-point subscales that tap the various domains of asthma management, with higher scores indicating better management (1 being the worse asthma management and 9 being the best asthma management). Mean of all of the subscales used to compute a total score.
Time Frame: 4 months from baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | 1: Home-based Family Intervention | 2: Enhanced Treatment As Usual
Number analyzed (Participants) | 21 | 20
units on a scale | 4.9 (.293) | 4.1 (.300)
Statistical Analysis 1: Comparison: 1: Home-based Family Intervention vs 2: Enhanced Treatment As Usual; Test type: Superiority or Other; p = 0.23, Regression, Linear — For both baseline to 4 month analyses (see above p value) and baseline to 10 month analyses, the variable of intervention group did not contribute significant additional variance; regression coefficient = .33

2. Primary Outcome: Metered Dose Inhaler Checklist (MDIC)
Description: Observational rating scale assessing MDI/spacer technique
Time Frame: 4 months, 10 months
Reporting Status: Not Posted

3. Primary Outcome: Asthma Morbidity, as Determined by Number of Asthma Symptom Days, Number of School Days Missed Due to Asthma, and Number of Emergency Department Visits for Acute Asthma
Time Frame: 4 months, 10 months
Reporting Status: Not Posted

4. Secondary Outcome: Parenting Stress Index - SF (PSI-SF)
Time Frame: 4 months, 10 months
Reporting Status: Not Posted

5. Secondary Outcome: Brief Symptom Inventory (BSI)
Time Frame: 4 months, 10 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 1: Home-based Family Intervention | 2: Enhanced Treatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes